CLINICAL TRIAL: NCT07290140
Title: A Randomized, Controlled, Blinded, Multi-Center Trial to Assess the Safety and Efficacy of Paclitaxel-Coated Sinus Balloon as an Adjunct to Endoscopic Sinus Surgery in Adult Chronic Rhinosinusitis Subjects
Brief Title: Paclitaxel-Coated Balloon Treatment of Chronic Rhinosinusitis
Acronym: RESTORE2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Airiver Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR3056
Record Dates: First submitted 2025-12-08; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Rhinosinusitis (CRS) With and Without Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- • Treatment with the Airiver ESSpand DCB and ESS (Experimental): Subjects will have ESSpand DCB dilation of the ESS treated sinuses
- Treatment with ESS (Active Comparator): Subjects will have ESS treatment at target sinuses
  Interventions: Procedure: ESS

INTERVENTIONS:
Combination Product: Airiver ESSpand DCB — The investigational procedure will be ESSpand DCB dilation of all surgically treated sinuses, including the resected ethmoid sinus cavities.
  Note: Prior to randomization to the investigational procedure, all subjects will undergo traditional ESS of their diseased sinuses.
Procedure: ESS — traditional ESS treatment of diseased sinuses.
  Arms: Treatment with ESS

SUMMARY:
This is a prospective, multicenter, randomized, controlled, double-blind clinical trial enrolling 300 adult subjects with chronic rhinosinusitis (CRS) with and without nasal polyps (CRSwNP and CRSsNP) indicated for endoscopic sinus surgery (ESS).

DETAILED DESCRIPTION:
Subjects will be randomized in a 1:1 ratio for ESS with no additional treatment (control group) or ESS followed by Airiver ESSpand DCB sinus dilation of affected sinuses (treatment group) at up to 40 US based sites.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years
2. Confirmed diagnosis of CRS per the 2021 "International Consensus Statement on Allergy and Rhinology: Rhinosinusitis" definition.
3. Radiographic evidence of bilateral ethmoid disease on CT taken 6 months or less prior to study index procedure and at least 6 months after any prior ESS or nasal surgery, polypectomy, balloon sinus dilation, etc. as applicable
4. Radiographic evidence of bilateral frontal sinus and/or frontal sinus outflow tract disease
5. Baseline SNOT-22 score ≥ 30
6. Has failed previous medical treatment and is an appropriate candidate for primary or revision ESS of bilateral ethmoid sinuses and bilateral frontal/frontal sinus outflow tract
7. Willing and able to provide written informed consent
8. Willing and able to comply with all protocol follow up visits and assessments

Exclusion Criteria:

1. Nasal cavity tumor (malignant or benign)
2. Antrochoanal polyps
3. Previous complete middle turbinate resection
4. Clinical evidence or suspicion of invasive fungal sinusitis (e.g., bone erosion on CT scan, necrotic sinus tissue)
5. History of prior lamina dehiscence or cerebrospinal fluid (CSF) leak in skull-based dehiscence
6. Concurrent condition requiring active chemotherapy and/or immunotherapy management
7. Subjects whose symptoms are too severe to undergo ESS (e.g., temperature >102.5F or extra-sinus manifestations, such as orbital cellulitis; dental or facial or brain abscess; cavernous vein thrombosis; or altered mental status
8. History of complications from prior ESS or balloon dilation procedure (e.g., CSF leak or injury to the skull base or orbital injury)
9. History of primary ciliary dyskinesia
10. Oral-steroid dependent conditions such as chronic obstructive pulmonary disease (COPD) or other conditions
11. Have evidence of significant baseline mucosal injury, ulceration, or erosion (e.g., exposed cartilage, perforation) on nasal examination
12. Acute purulent nasal infection or upper respiratory tract infection, including but not limited to acute bacterial rhinosinusitis (ABRS), acute rhinosinusitis (ARS), or COVID -19 within 2 weeks before the baseline visit.
13. Allergy or hypersensitivity to paclitaxel or structurally related compounds.
14. Subject has taken biologic drugs in the 6 months leading up to the screening visit or who expect to take biologics in the next 24 months.
15. Subject has taken oral corticosteroids in the 30 days leading up to their baseline appointment.
16. Subject who plans to undergo posterior nasal nerve ablation in the next 24 months.
17. Subject has a history of inability to tolerate nasal endoscopy
18. Concurrent medical condition that would affect the investigator's ability to evaluate the subject's condition or that could compromise subject safety, such as severe COPD, severe asthma
19. Pregnant or planning to become pregnant during the first 12 months of enrollment in the study
20. Subject who has undergone a nasal/sinus surgery including but not limited to ESS, polypectomy, septoplasty, turbinoplasty, balloon sinus dilation, placement of steroid releasing implants, posterior nasal nerve ablation in the 6 months prior to the baseline appointment.
21. Previous Draf III frontal sinus surgery or a study index procedure ESS is expected to be or is a Draf III sinus surgery.
22. Subject whose index procedure did not include bilateral ethmoid ESS and bilateral frontal ESS
23. Subject whose expected study index procedure includes steroid releasing implants or non-resorbable nasal packing/stents.
24. Subject whose study index procedure is aborted for any reason
25. Life expectancy <2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-28 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary safety | 30 days post- index procedure
  Incidence of major adverse events (MAE) through 30 days post-index treatment.
Primary efficacy endpoint | 6 months post-index procedure
  Reduction in need for postoperative intervention in the ethmoid and /or frontal sinus within 6 months post-index procedure.

SECONDARY OUTCOMES:
Hypothesis tested clinical responder rate at 12 months | 12 months
  a responder is defined as a subject who has not undergone revision ESS, balloon sinus dilation, or any other procedural intervention, or received oral/systemic steroid or biologic therapy for CRS in the follow-up period, and with SNOT-22 score change from baseline (CFBL) by ≥8.9 points
Hypothesis tested mean adhesion/scaring grade of sphenoid sinus at 6 months, as assessed by the independent, blinded reviewer | 6 months
  Grading 0 to 3, the higher grade indicates significant scarring and adhesion

CONTACTS AND LOCATIONS:
Overall Officials: Noem Cohen, MD, Principal Investigator — University of Pennsylvania; Rodney Schlosser, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Airiver Medical, Brooklyn Park, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided